CLINICAL TRIAL: NCT03736447
Title: Peanut Oral Immunotherapy Study of Early Intervention for Desensitization (POSEIDON)
Brief Title: Peanut Oral Immunotherapy Study of Early Intervention for Desensitization
Acronym: POSEIDON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARC005
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Results first posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Peanut Allergy
Keywords: CODIT™ (characterized oral desensitization immunotherapy™); Peanut-Allergic Children; CPNA (Characterized Peanut Allergen); Desensitization; AR101; Allergy; Peanut Allergy; Characterized Peanut Allergen; Oral Immunotherapy
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity | interventions — Capsules

STUDY DESIGN:
Intervention Model Description: 2:1 randomization
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AR101 powder provided in capsules & sachets (Active Comparator): Study product provided as peanut protein in pull-apart capsules or sachets
  Interventions: Biological: AR101 powder provided in capsules & sachets
- Placebo powder provided in capsules & sachets (Placebo Comparator): Placebo formulation in pull-apart capsules or sachets containing only inactive ingredients
  Interventions: Biological: Placebo powder provided in capsules & sachets

INTERVENTIONS:
Biological: AR101 powder provided in capsules & sachets — Study product formulated to contain peanut protein at different dosage strengths for use as defined in the protocol
  Arms: AR101 powder provided in capsules & sachets
Biological: Placebo powder provided in capsules & sachets — Study product formulated to contain only inactive ingredients for use as defined in the protocol
  Arms: Placebo powder provided in capsules & sachets

SUMMARY:
The purpose of this study is to determine the efficacy and safety of AR101 in peanut-allergic children aged 1 to < 4 years.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled study conducted at 14 study sites in North America and 9 in Europe to evaluate the efficacy and safety of AR101 in a characterized oral desensitization immunotherapy (CODIT™) regimen compared with placebo in peanut-allergic children aged 1 to < 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 to < 4 years at randomization.
* Written informed consent from the legal guardian/parent (or both parents where required by local authorities). Provide assent where required and as appropriate per local requirements.
* Sensitivity to peanut, defined as one of the following:

  * No known history of peanut ingestion and has serum IgE to peanut ≥ 5 kUA/L within 12 months before randomization.
  * Documented history of physician-diagnosed IgE-mediated peanut allergy that includes the onset of characteristic* signs and symptoms of allergy within 2 hours of known oral exposure to peanut or peanut-containing food, and has a mean wheal diameter on skin prick test (SPT) to peanut of at least 3 mm greater than the negative control (diluent) or serum IgE to peanut ≥ 0.35 kUA/L, obtained within 12 months before randomization.
* Development of age-appropriate dose-limiting allergy symptoms after consuming single doses of peanut protein > 3 mg to ≤ 300 mg in a screening DBPCFC.
* A palatable vehicle food to which the subject is not allergic must be available for administering study product.

Exclusion Criteria:

* History of severe or life-threatening anaphylaxis anytime before the screening DBPCFC.
* History of hemodynamically significant cardiovascular or renovascular disease, including uncontrolled or inadequately controlled hypertension.
* History of biopsy-confirmed diagnosis of EoE; other eosinophilic GI disease; chronic, recurrent, or severe gastroesophageal reflux disease (GERD); or symptoms of dysphagia (eg, difficulty swallowing, food "getting stuck").
* Recurrent GI symptoms considered clinically significant in the opinion of the investigator.
* History of a mast cell disorder including mastocytosis, urticaria pigmentosa, chronic idiopathic or chronic physical urticaria beyond simple dermatographism (eg, cold urticaria, cholinergic urticaria), and hereditary or idiopathic angioedema.
* Moderate or severe persistent asthma (criteria steps 3-6; National Heart, Lung, and Blood Institute [NHLBI], 2007).
* Mild asthma (criteria steps 1-2; NHLBI, 2007) that is uncontrolled or difficult to control based on NHLBI 2007 criteria.
* History of high-dose corticosteroid use (eg, 1-2 mg/kg prednisone or equivalent for > 3 days) by any route of administration as defined by any of the following:

  * Steroid administered daily for > 1 month within 1 year before screening
  * One steroid course within 6 months before screening
  * More than 2 steroid courses ≥ 1 week in duration within 1 year before screening
* History of food protein-induced enterocolitis syndrome (FPIES) within 12 months before screening.
* Recurrent urticaria.
* History of failure to thrive or any other form of abnormal growth, or developmental or speech delay that precludes age-appropriate communication.
* History of chronic disease (except mild intermittent asthma, mild persistent asthma that is controlled, atopic dermatitis, or allergic rhinitis) that is or is at significant risk of becoming unstable or requiring a change in a chronic therapeutic regimen.
* Unable to discontinue antihistamines and other medications that could interfere with the assessment of an allergic reaction for 5 half-lives of the medication before the screening SPT, first day of dose escalation, and DBPCFCs.
* Use or anticipated use of a prohibited medication (eg, beta blockers [oral], angiotensin converting enzyme inhibitors, angiotensin receptor blockers, calcium channel blockers, or tricyclic antidepressants), monoclonal antibody, or any other immunomodulatory therapy (including immunosuppressive medications).
* Treatment with any form of immunotherapy for any food allergy anytime before screening.
* Participation in another clinical trial within 30 days or 5 half-lives of the investigational product, whichever is longer, before screening.
* Allergy to oat or rice.
* Hypersensitivity to epinephrine or any of the excipients in the epinephrine auto-injector.
* Parent/caregiver unable or unwilling to use epinephrine auto-injectors.
* Unable to follow the protocol requirements.
* Any other condition (concurrent disease, infection, comorbidity, or psychiatric or psychological disorders) or reason that may interfere with the ability to participate in the study, cause undue risk, or complicate the interpretation of data, in the opinion of the investigator or medical monitor.
* Resides at the same place as another subject in any AR101 interventional trial.
* Lives in the same household and/or is a family member of a sponsor employee or site staff involved in conducting this study.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Director — Aimmune Therapeutics
Locations (23):
- United States (14):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Sean N. Parker Center for Allergy & Asthma Reseach, LPCH at El Camino Hospital, Mountain View, California
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - Allergy & Asthma Medical Group and Research Center, San Diego, California
  - Children's Center for Advanced Pediatrics Clinical Research Lab, Atlanta, Georgia
  - Atlanta Allergy & Asthma Clinic, Marietta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The John Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Division of Allergy and Clinical Immunology, Ann Arbor, Michigan
  - Atlantic Research Center, Ocean City, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UNC-CH School of Medicine, Pediatric Allergy, Immunology & Rheumatology, Food Allergy, Chapel Hill, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Virginia Mason Medical Center, Seattle, Washington
- Jeanne de Flandre Hospital, Lille, France
- Germany (2):
  - Charité Universitaetsmedizin Berlin, Berlin
  - University of Frankfurt, Frankfurt am Main
- United Kingdom (6):
  - James Paget University Hospital, Gorleston-on-Sea, Norfolk
  - Leicester Royal Infirmary, Leicester
  - Guy's and St. Thomas' NHS Foundation Trust, Snowy Owl, First Floor, Evelina Children's Hospital, London
  - Royal Manchester Children's Hospital Central Manchester University Hospitals, Manchester
  - Sheffield Children's Hospital, Sheffield
  - University Hospital Southampton Foundation NHS Trust Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Du Toit G, Brown KR, Vereda A, Irani AM, Tilles S, Ratnayake A, Jones SM, Vickery BP. Oral Immunotherapy for Peanut Allergy in Children 1 to Less Than 4 Years of Age. NEJM Evid. 2023 Nov;2(11):EVIDoa2300145. doi: 10.1056/EVIDoa2300145. Epub 2023 Oct 23. PMID 38320526

RESULTS

PARTICIPANT FLOW:
Groups:
- AR101: AR101 drug product was supplied in 2 presentations. These were pull-apart capsules containing 0.5, 1, 10, 20 and 100mg of peanut protein and sealed, foil-laminated sachets containing 300mg of peanut protein. Contents were delivered over an age-appropriate semisolid, vehicle food and mixed thoroughly.
  The capsules were used during the Initial Escalation and Up-dosing phases of the study. The sachets were used during the Maintenance phase.
- Placebo: A Placebo matching the AR101 drug product was supplied in 2 presentations. These were pull-apart capsules matching the 0.5, 1, 10, 20 and 100mg peanut capsules but containing no peanut protein, and sealed, foil-laminated sachets matching the peanut protein sachets but without any peanut protein. Contents were delivered over an age-appropriate semisolid, vehicle food and mixed thoroughly.
  The capsules were used during the Initial Escalation and Up-dosing phases of the study. The sachets were used during the Maintenance phase.
Period: Overall Study
Arm/Group | AR101 | Placebo
Started | 98 | 48
Completed | 83 | 45
Not Completed | 15 | 3
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Continued commitment to study treatment | 3 | 0
Not completed — Taste aversion to study product | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AR101 | Placebo | Total
Number analyzed (Participants) | 98 | 48 | 146
Age, Customized [Count of Participants; unit: Participants]
  1-<2 years | 33 | 16 | 49
  2-<3 years | 35 | 15 | 50
  3-<4 years | 30 | 17 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 20 | 61
  Male | 57 | 28 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 75 | 31 | 106
  Unknown or Not Reported | 18 | 14 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 8 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 65 | 28 | 93
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Tolerated a Single Highest Dose of at Least 600 mg in the Exit Double-Blind, Placebo-Controlled Food Challenge (DBPCFC)
Description: The percentage of subjects in the ITT population who achieve desensitization as determined by tolerating specified challenge doses of peanut protein with no more than mild allergy symptoms during the exit double-blind placebo-controlled food challenge (DBPCFC).
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 98 | 48
Percentage of subjects | 73.5 [63.6 to 81.9] | 6.3 [1.3 to 17.2]
Statistical Analysis 1: Comparison: AR101 vs Placebo; Test type: Superiority; p < 0.0001, Farrington-Manning test; Risk Difference (RD) = 67.2, 95% CI 2-sided [50.0 to 84.5]

2. Secondary Outcome: Percentage of Subjects Who Tolerated a Single Highest Dose of at Least 1000 mg in the Exit Double-Blind, Placebo-Controlled Food Challenge (DBPCFC) [Time Frame: 12 Months]
Description: as for outcome 1
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 98 | 46
Percent of participants | 68.4 [58.2 to 77.4] | 4.2 [0.5 to 14.3]
Statistical Analysis 1: Comparison: AR101 vs Placebo; Test type: Superiority; p < 0.0001, Farrington-Manning test; Risk Difference (RD) = 64.2, 95% CI 2-sided [47.0 to 81.4]

3. Secondary Outcome: Percentage of Subjects Who Tolerated a Single Highest Dose of at Least 300 mg in the Exit Double-Blind, Placebo-Controlled Food Challenge (DBPCFC)
Description: as for outcome 1
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 98 | 48
Percentage of subjects | 79.6 [70.3 to 87.1] | 22.9 [12.0 to 37.3]
Statistical Analysis 1: Comparison: AR101 vs Placebo; Test type: Superiority; p < 0.0001, Farrington-Manning test; Risk Difference (RD) = 56.7, 95% CI 2-sided [39.8 to 73.5]

4. Secondary Outcome: Maximum Severity of Symptoms in Participants at Any Challenge Dose During the Exit Double-blind Placebo Controlled Food Challenge (DBPCFC)
Description: The maximum severity of symptoms that occurred at any challenge dose of peanut protein during the exit DBPCFC.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 98 | 48
Participants
  None | 50 | 2
  Mild | 29 | 23
  Moderate | 17 | 21
  Severe | 2 | 2
  Life-threatening or fatal | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | AR101 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/48
Serious Adverse Events (participants affected / at risk) | 7/98 | 2/48
Other Adverse Events (participants affected / at risk) | 96/98 | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR101 (N=98) | Placebo (N=48)
Enterovirus infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Status asthmaticus (Infections and infestations) | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR101 (N=98) | Placebo (N=48)
Vomiting (Gastrointestinal disorders) | 52 | 15
Diarrhoea (Gastrointestinal disorders) | 34 | 13
Abdominal pain (Gastrointestinal disorders) | 23 | 6
Abdominal pain upper (Gastrointestinal disorders) | 14 | 4
Constipation (Gastrointestinal disorders) | 11 | 5
Oral pruritus (Gastrointestinal disorders) | 10 | 2
Teething (Gastrointestinal disorders) | 10 | 7
Flatulence (Gastrointestinal disorders) | 5 | 0
Lip swelling (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 35 | 13
Nasopharyngitis (Infections and infestations) | 28 | 13
Rhinitis (Infections and infestations) | 20 | 8
Ear infection (Infections and infestations) | 11 | 2
Gastroenteritis (Infections and infestations) | 10 | 6
Viral infection (Infections and infestations) | 9 | 5
Viral upper respiratory tract infection (Infections and infestations) | 9 | 5
Gastroenteritis viral (Infections and infestations) | 8 | 1
Conjunctivitis (Infections and infestations) | 6 | 5
Corona virus infection (Infections and infestations) | 6 | 6
Hand-foot-and-mouth disease (Infections and infestations) | 5 | 2
Influenza (Infections and infestations) | 5 | 0
Lower respiratory tract infection (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 5 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 51 | 24
Erythema (Skin and subcutaneous tissue disorders) | 34 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 15
Eczema (Skin and subcutaneous tissue disorders) | 24 | 12
Rash (Skin and subcutaneous tissue disorders) | 23 | 11
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 17 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 8 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 | 5
Swelling face (Skin and subcutaneous tissue disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 21
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 42 | 15
Sneezing (Respiratory, thoracic and mediastinal disorders) | 23 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 14 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pyrexia (General disorders) | 50 | 20
Arthropod bite (Injury, poisoning and procedural complications) | 7 | 2
Head injury (Injury, poisoning and procedural complications) | 6 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 0
Eye pruritus (Eye disorders) | 9 | 5
Eye swelling (Eye disorders) | 9 | 3
Ocular hyperaemia (Eye disorders) | 6 | 2
Anaphylactic reaction (Immune system disorders) | 8 | 4
Seasonal allergy (Immune system disorders) | 4 | 4
Headache (Nervous system disorders) | 10 | 1
Irritability (Psychiatric disorders) | 6 | 1
Ear pain (Ear and labyrinth disorders) | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT03736447/Prot_SAP_000.pdf